CLINICAL TRIAL: NCT02776696
Title: Comparison of Two Closed-Loop Strategies for Glucose Control in Type 1 Diabetes The DREMED Trail- 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: rmc082315ctil
Record Dates: First submitted 2016-05-16; First posted 2016-05-18 (Estimated); Last update posted 2019-12-27 (Actual); Status verified 2018-09

CONDITIONS: Type 1 Diabetes
Keywords: Closed Loop; Artificial Pancreas
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: segment 1 part 1 is a single arm study, segment 1 part 2 is a is a crossover study, segment 2 is a randomized crossover study , segment 3 is a parallel study and segment 4 is a single arm study
Oversight: Data Monitoring Committee: No

ARMS (2):
- Advanced HybridClosed Loop System (AHCL) (Experimental): Advanced Hybrid Closed Loop System (AHCL) - all subjects wearing the study system during 36 hours in the clinic during segment 1or 2 days in a camp setting during segment 2 or 12 days in a camp setting during segment 3 or 5 days in a camp setting and 21 days at home during segment 4.
  Interventions: Device: Advanced Hybrid Closed Loop System
- Hybrid Closed Loop System (HCL) (Experimental): Hybrid Closed Loop System (HCL) - all subjects wearing the study system during:
  36 hours in the clinic during segment 1or 2 days in a camp setting during segment 2 or 12 days in a camp setting during segment 3
  Interventions: Device: Hybrid Closed Loop System

INTERVENTIONS:
Device: Advanced Hybrid Closed Loop System
  Other Names: AHCL
  Arms: Advanced HybridClosed Loop System (AHCL)
Device: Hybrid Closed Loop System
  Other Names: HCL
  Arms: Hybrid Closed Loop System (HCL)

SUMMARY:
The purpose of the study is to compare two closed-loop strategies in terms of glycemic control in Type 1 Diabetes during a camp setting.

The proposed study is a four-segment feasibility study. One segment is a proof of concept study (with two parts) conducted as in-patient clinic study ,the second segment is two-arms, cross-over, randomized and single-center and the third segment is four-arms, parallel, randomized and single-center, in diabetes camp study in subjects with type 1 diabetes on insulin pump therapy and the forth segment is a single arm feasibility in a diabetes camp setting followed by a 3 weeks period at home.

Segment 1 will be divided into two parts: part 1 is a single arm pilot study aim to asses logistical and safety issues in 12 patients and part 2 is a randomized cross over study aim to evaluate glucose performance using closed-loop control. Part 2-is a randomized cross-over (two arms) in-patient study: A total of 12 patients will participate in this part of the study. Following the run-in period subjects will be randomized to participate in two periods of closed-loop treatment, each period will last 36 hours in hospital setting. During the first period, glycemic control will be controlled by the Hybrid closed-loop system and during the second period by Hybrid Logic closed-loop system. The sequence of treatment first period HCL therapy than AHCL or vice versa will be randomly assigned.

Segment 2 is a randomized cross-over (two arms) Camp Study including up to 30 patients. Following the run-in period subjects will be randomized to participate in two periods of closed-loop treatment, each period will last 2days in a camp setting, the total duration of the camp will be up to 6 days. In one period, glycemic control will be controlled by the Hybrid closed-loop system and another period by Hybrid Logic closed-loop system. The sequence of treatment first period HCL therapy than AHCL or vice versa will be randomly assigned.

Segment 3 is a randomized, parallel (four arm) Camp Study including up to 80 patients. Following the run-in period subjects will be randomized to participate in one of 4 intervention arms of closed-loop treatment in camp settings. The duration of the camp will be 12 days in which glycemic control will be controlled by one of 4 versions of closed-loop system: Hybrid Closed Loop (HCL) or one of 3 versions of Advanced Hybrid Closed Loop (AHCL).

Segment 4 is a single arm, feasibility study in a diabetes camp setting followed by a three week period at home. After the completion of segments 1-3, the AHCL system will be optimized and a new version of the system will be created for use in segment 4. Up to 20 subjects will participate in this part of the study. Following a minimum of 5 days run-in period, subjects will be placed in a camp setting and closed loop will be initiated. Subjects will remain in closed loop for 5 days and will have 3 days of challenges, including missed meal bolus, late meal bolus and moderate-intensity exercise. At the conclusion of the camp, subjects will continue to use the system at home in Auto Mode for a period of 21 days.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes duration > 1 year since diagnosis
* Pump therapy for at least 6 months and experience with sensor use
* Age10-40 years: Age 10-30 for segments 1-3, Age 14-40 for segment 4.
* 7>HbA1c <10.0 at time of screening visit for segments 1 and 2, <10.0 at segments 3 and 4.
* Willing to follow study instructions
* Willing to perform ≥ 3 finger stick blood glucose measurements daily
* Willing to perform required sensor calibrations
* Patient capable of reading and understand instructions in English
* Willing to have an adult experienced in the management of diabetes to live with during the outpatient phase of the protocol.

Exclusion Criteria:

* Subject is unable to tolerate tape adhesive in the area of sensor placement
* Subject has any unresolved adverse skin condition in the area of sensor or device placement
* Subject is actively participating in an investigational study (drug or device) wherein they have received treatment from an investigational study (drug or device) in the last 2 weeks
* Subject has a positive pregnancy screening test
* Subject is female, sexually active without the use of contraception, and plans/able to become pregnant during the course of the study and is not using an acceptable method of contraception
* Subject has had a hypoglycemic seizure within the past 6 months prior to screening visit
* Subject has had hypoglycemia resulting in loss of consciousness within the past 6 months prior to screening visit
* Subject has had an episode of diabetic ketoacidosis (DKA) within the past 6 months prior to screening visit
* Subject has a history of a seizure disorder
* Subject has central nervous system or cardiac disorder resulting in syncope
* Subject has a history of myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack (TIA), cerebrovascular accident (CVA), angina, congestive heart failure, ventricular rhythm disturbances or thromboembolic disease
* Subjects with hematocrit lower than the normal reference range per local lab testing
* Subjects with a history or findings on screening electrocardiogram of any cardiac arrhythmia
* Subjects with a history of adrenal insufficiency
* Subjects with history of migraines that have occurred at least 2 times in the last 3 months prior to enrollment
* Any disease or condition that may influence the HbA1c testing
* Subject needs to travel by air during the study duration.

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2016-06; Primary Completion 2019-08-14 (Actual); Study Completion 2019-08-14 (Actual)

PRIMARY OUTCOMES:
Percentage of glucose sensor readings within 70 to 180 mg/dl | Day 21 for segments 1-3 , day 5 for segment 4 camp portion and day 31 for segment 4 home portion

SECONDARY OUTCOMES:
Area Under the Curve of glucose sensor readings below 70 mg/dl | Day 21 for segments 1-3 , day 5 for segment 4 camp portion and day 31 for segment 4 home portion
Percentage of glucose sensor readings below 70 mg/dl | Day 21 for segments 1-3 , day 5 for segment 4 camp portion and day 31 for segment 4 home portion
Area Under the Curve of glucose sensor readings above 180 mg/dl | Day 21 for segments 1-3 and day 31 for segment 4
Percentage of glucose sensor readings above 180 mg/dl | Day 20
Average of glucose sensor readings | Day 21 for segments 1-3 , day 5 for segment 4 camp portion and day 31 for segment 4 home portion
Standard Deviation of glucose sensor readings | Day 21 for segments 1-3 , day 5 for segment 4 camp portion and day 31 for segment 4 home portion
Time in glucose range of 70-180 mg/dl during day time (6am-12am) | Day 21 for segments 1-3 , day 5 for segment 4 camp portion and day 31 for segment 4 home portion
Time in glucose range of 70-180 mg/dl during night time (12am-6am) | Day 21 for segments 1-3 , day 5 for segment 4 camp portion and day 31 for segment 4 home portion
Area Under the Curve of glucose sensor readings above 250 mg/dL | Day 21 for segments 1-3 , day 5 for segment 4 camp portion and day 31 for segment 4 home portion
Area Under the Curve of glucose sensor readings above 300 mg/dL | Day 21 for segments 1-3 , day 5 for segment 4 camp portion and day 31 for segment 4 home portion
Percentage of glucose sensor readings above 250 mg/dL | Day 21 for segments 1-3 , day 5 for segment 4 camp portion and day 31 for segment 4 home portion
Percentage of glucose sensor readings above 300 mg/dL | Day 21 for segments 1-3 , day 5 for segment 4 camp portion and day 31 for segment 4 home portion
Area Under the Curve of glucose sensor readings below 50 mg/dL | Day 21 for segments 1-3 , day 5 for segment 4 camp portion and day 31 for segment 4 home portion
Area Under the Curve of glucose sensor readings below 60 mg/dL | Day 21 for segments 1-3 , day 5 for segment 4 camp portion and day 31 for segment 4 home portion
Percentage of glucose sensor readings below 50 mg/dL | Day 21 for segments 1-3 , day 5 for segment 4 camp portion and day 31 for segment 4 home portion
Percentage of glucose sensor readings below 60 mg/dL | Day 21 for segments 1-3 , day 5 for segment 4 camp portion and day 31 for segment 4 home portion
Percentage of time in Closed Loop | Day 21 for segments 1-3 , day 5 for segment 4 camp portion and day 31 for segment 4 home portion
Sensor mean absolute relative difference (MARD) | Day 21 for segments 1-3 , day 5 for segment 4 camp portion and day 31 for segment 4 home portion
Total insulin dose | Day 21 for segments 1-3 , day 5 for segment 4 camp portion and day 31 for segment 4 home portion
Serious Adverse Events (SAE) | Day 21 for segments 1-3 , day 5 for segment 4 camp portion and day 31 for segment 4 home portion
Serious Adverse Device Events (SADE) | Day 21 for segments 1-3 , day 5 for segment 4 camp portion and day 31 for segment 4 home portion
Unanticipated Adverse Device Effects (UADE) | Day 21 for segments 1-3 , day 5 for segment 4 camp portion and day 31 for segment 4 home portion
Incidence of Severe Hypoglycemia | Day 21 for segments 1-3 , day 5 for segment 4 camp portion and day 31 for segment 4 home portion
Incidence of Diabetic Ketoacidosis (DKA) | Day 21 for segments 1-3 , day 5 for segment 4 camp portion and day 31 for segment 4 home portion
Closed-loop acceptance questionnaire | Day 21 for segments 1-3 , day 5 for segment 4 camp portion and day 31 for segment 4 home portion
  The questionnaire contains 5 sections evaluating the user acceptance of the study devise (general satisfaction, comparison to previous treatment, importance of the system, expectations from the system and suggestions for improvement) each section consists of 1-31 questions each, with specific scales for each of the questions. Subscales are not combined to compute a total score.

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, Prof, Principal Investigator — Schneider Children's Medical Center
Locations (1):
- Schneider Children's Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No